CLINICAL TRIAL: NCT05526222
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study of Jaktinib Hydrochloride Tablets in the Treatment of Adult Patients With Moderate and Severe Atopic Dermatitis
Brief Title: A Phase III Study of Jaktinib in Adults With Moderate and Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZGJAK025
Record Dates: First submitted 2022-08-25; First posted 2022-09-02 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jaktinib low dose (Experimental): Low dose
  Interventions: Drug: Jaktinib Hydrochloride Tablet
- Jaktinib high dose (Experimental): High dose
  Interventions: Drug: Jaktinib Hydrochloride Tablet
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Jaktinib Hydrochloride Tablet

INTERVENTIONS:
Drug: Jaktinib Hydrochloride Tablet — Orally administered, twice a day

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled phase III clinical study of jaktinib hydrochloride tablets in the treatment of adult patients with moderate and severe atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Have fully understood the test and voluntarily signed the informed consent;
* When signing the informed consent form, the age of male or female subjects must be ≥ 18 years old;
* The onset time of atopic dermatitis was at least 1 year at the time of screening, and the subjects met the Hanifin and Rajka criteria for atopic dermatitis at the time of screening;
* For women with reproductive ability and all male subjects, during the trial period and within 6 months after the discontinuation of the trial drug, they must maintain abstinence or contraception, including but not limited to physical and drug contraception.
* The subjects were able to communicate well and agreed to follow the study and follow-up procedures.

Exclusion Criteria:

* The investigator considers that any subjects are not suitable to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The efficacy in the treatment of moderate and severe atopic dermatitis | 16 weeks
  The proportion of subjects whose Eczema Area and Severity Index (EASI) total score decreased by ≥ 75% from baseline
The efficacy in the treatment of moderate and severe atopic dermatitis | 16 weeks
  The proportion of subjects with a systemic Investigator's Global Assessment (IGA) score of 0 or 1 and a decrease of ≥ 2 points from baseline

SECONDARY OUTCOMES:
The abnormal laboratory values and/or adverse events in the treatment of moderate and severe atopic dermatitis | up to 1 year
  Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Director — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- 139 People's Middle Road, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No